CLINICAL TRIAL: NCT01280266
Title: Comparison of Phosphodiesterase-5 Inhibitor and Calcium Channel Inhibitor for the Treatment of Secondary Raynaud Phenomenon, Double Blind, Randomized, Cross-over Trial
Brief Title: Efficacy Study of PDE-5 Inhibitor and Calcium Channel Inhibitor for the Treatment of Secondary Raynaud Phenomenon
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Eun Bong Lee, Direct, Division of Rheumatology, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RaynaudSNUH
Record Dates: First submitted 2011-01-14; First posted 2011-01-20 (Estimated); Results first posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Raynaud Phenomenon
Keywords: Pathological Conditions; Signs and Symptoms; Blood circulation
MeSH Terms: conditions — Raynaud Disease; Signs and Symptoms | interventions — udenafil; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Amlodipine-Udenafil (AU) arm (Experimental): Amlodipine 10mg PO QD for 4 weeks, washout period, then Udenafil 100mg PO QD for 4 weeks
  Interventions: Drug: Udenafil or Amlodipine
- Udenafil-Amlodipine (UA) arm (Experimental): Udenafil 100mg PO QD for 4 weeks, washout period, then Amlodipine 10mg PO QD for 4 weeks
  Interventions: Drug: Udenafil or Amlodipine

INTERVENTIONS:
Drug: Udenafil or Amlodipine — Amlodipine 10mg daily then Udenafil 100 mg daily OR Udenafil 100 mg daily then Amlodipine 10mg daily

SUMMARY:
The prevalence of Raynaud phenomenon (RP), a reversible vaso-constriction with skin discoloration, is 5-10% in general population. Often conventional measures such as warming up or minimizing exposure to cold are not enough and many patients require treatment with a vasodilator therapy. A recent study showed a good efficacy and safety profile of sildenafil, a selective inhibitor of cGMP specific phosphodiesterase type 5 (PDE5) in RP.

Here, the investigators aim to examine the efficacy and safety of Udenafil, a newer PDE5 inhibitor, as compared to amlodipine, a well known calcium channel blocker, in the treatment of secondary RP in Korean patients.

ELIGIBILITY:
Inclusion Criteria:

* secondary Raynaud's phenomenon

Exclusion Criteria:

* primary raynaud phenomenon
* active infection
* hypersensitivity to PDE5 inhibitor or Calcium Chanel Blocker (CCB)
* elevated AST/ALT (3 times above the upper normal limit)
* severe renal failure
* patients on nitrite or nitric oxide (NO) donor treatment
* recent history of cerebrovascular accidents, acute myocardial infarction, or coronary artery bypass surgery
* hypotension (less than 90/50 mmHg) or uncontrolled hypertension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eun Bong Lee, MD PhD, Principal Investigator — professor of Seoul National University College of Medicine; Eun Young Lee, MD PhD, Study Director — Assistant professor, Seoul National University College of Medicine; Jin Kyun Park, MD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee EY, Park JK, Lee W, Kim YK, Park CS, Giles JT, Park JW, Shin K, Lee JS, Song YW, Lee EB. Head-to-head comparison of udenafil vs amlodipine in the treatment of secondary Raynaud's phenomenon: a double-blind, randomized, cross-over study. Rheumatology (Oxford). 2014 Apr;53(4):658-64. doi: 10.1093/rheumatology/ket417. Epub 2013 Dec 17. PMID 24352340

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment begin Jan 13 2011 until Mar 15 2011. Location: Rheumatology outpatient clinic at Seoul National University Hospital, Seoul, Korea.
Pre-assignment Details: 30 Patients were initially recruited, but an error occurred in obtaining informed consent and this one was withdrawn.
Groups:
- Amlodipine-Udenafil (AU) Arm: Amlodipine 10mg PO QD for 4 weeks, washout period for 1week, then Udenafil 100mg PO QD for 4 weeks.
- Udenafil-Amlodipine (UA) Arm: Udenafil 100mg PO QD for 4 weeks, washout period for 1 week, then Udenafil 10mg PO QD for 4 weeks.
Period: First Intervention (Week 1-4)
Arm/Group | Amlodipine-Udenafil (AU) Arm | Udenafil-Amlodipine (UA) Arm
Started | 15 | 14
Completed | 14 | 12
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Period: Washout Period (Week 4-5)
Arm/Group | Amlodipine-Udenafil (AU) Arm | Udenafil-Amlodipine (UA) Arm
Started | 14 | 12
Completed | 14 | 12
Not Completed | 0 | 0
Period: Second Intervention (Week 5-9)
Arm/Group | Amlodipine-Udenafil (AU) Arm | Udenafil-Amlodipine (UA) Arm
Started | 14 | 12
Completed | 14 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Amlodipine-Udenafil (AU) Arm: Amlodipine first, then Udenafil
- Udenafil-Amlodipine (UA) Arm: Udenafil first, then Amlodipine
- Total: Total of all reporting groups
Arm/Group | Amlodipine-Udenafil (AU) Arm | Udenafil-Amlodipine (UA) Arm | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 26
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49.6 (14.0) | 52.3 (10.3) | 50.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 14 | 12 | 26
Disease subtype [Number; unit: participant] — Underlying rheumatic disease
  participant
    Localized systemic sclerosis (SSc) | 1 | 2 | 3
    diffuse SSc | 10 | 7 | 17
    Mixed connective tissue disease | 1 | 2 | 3
    Sjogren's disease | 2 | 1 | 3
RP duration [Mean (Standard Deviation); unit: years] | 8.8 (8.7) | 5.6 (2.3) | 7.3 (6.6)
Prior use of vasodilator [Number; unit: Participant]
  calcium channel blocker | 1 | 4 | 5
  angiotensin receptor blocker | 2 | 0 | 2
  Pentyxifylline | 1 | 1 | 2
  No prior use | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: RP Attacks Per Day
Description: Change in RP frequency after amlodipine and udenafil number of RP attack per day 0 -- unlimited.
Time Frame: baselin and 4 weeks
Population: 14 patients in UA arm + 12 patients in AU arm
Measure: Mean (Standard Deviation); unit: attacks per day
Groups:
- Amlodipine: Changes in RP attacks per day during amlodipine 10 mg orally per day
- Udenafil: Changes in RP attacks per day during udenafil 100mg orally per day
Arm/Group | Amlodipine | Udenafil
Number analyzed (Participants) | 26 | 26
attacks per day | -0.5 (1.4) | -0.5 (0.9)

2. Secondary Outcome: Change in Raynaud's Condition Score (RCS)
Description: change in the RCS. RCS combines daily activty, frequency, duration and severity as well as impact of RP attack (Measuring disease activity and functional status in patients with scleroderma and Raynaud's phenomenon, Merkel et al,Arthritis Rheum. 2002 Sep;46(9):2410-20).
  Range 0-10 ordinal scale 0..good 10.. bad
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Amlodipine: Changes in RPS during amlodipine 100 mg orally per day
- Udenafil: Changes in RPS during udenafil 10 mg orally per day
Arm/Group | Amlodipine | Udenafil
Number analyzed (Participants) | 26 | 26
units on a scale | -0.5 (1.5) | -0.3 (1.0)

3. Secondary Outcome: Change in the RP Duration
Description: Change in the average RP duration in minutes (min) per attack. 0 -- unlimited
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: min per attack
Groups:
- Amlodipine: Drug: amlodipine 100 mg p.o. per day
- Udenafil: Drug: udenafil 10 mg p.o. per day
Arm/Group | Amlodipine | Udenafil
Number analyzed (Participants) | 26 | 26
min per attack | -1.1 (5.9) | -1.4 (11.4)

4. Secondary Outcome: Change in Health Assessment Questionnaire (HAQ)
Description: Ordinal scale 0-10 0 good 10 bad
Time Frame: 0 and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amlodipine | Udenafil
Number analyzed (Participants) | 26 | 26
units on a scale | 0.1 (0.4) | -0.1 (0.3)

5. Secondary Outcome: Change in Physician's Global Assessment on Visual Analogue Scale (VAS)
Description: Physician's global assessment (PGA) on VAS assesses the overall condition of the patient. The scale ranges from 0 - 10, with 0 being good and 10 bad. As such, change in the GPA measures the change in the patient's condition from the baseline.
  negative value (decrease in value) means improvement.
Time Frame: at 0 (baseline) and 4 weeks (after treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amlodipine | Udenafil
Number analyzed (Participants) | 26 | 26
units on a scale | -0.9 (1.4) | -1.5 (1.6)

6. Secondary Outcome: Change in Digital Ulcer Number
Description: 0 - unlimited. Number of digital ulcers in all fingers are counted by the investigators and recorded at each visit. The number of ulcers in all fingers indirectly reflect the extent of critical ischemia. As such. the decrease in digital ulcer number reflects positive response to treatment (=better blood flow), whereas the increase ulcer numbers indicates worsening finger ischemia from baseline.
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: Digital ulcers
Arm/Group | Amlodipine | Udenafil
Number analyzed (Participants) | 26 | 26
Digital ulcers | 0.1 (0.4) | 0.1 (0.3)

7. Secondary Outcome: Change in Peak Systolic Flow (cm/Sec)
Description: Change in digital artery flow velocity in proper palmar digital artery in cm/sec.
  0-unlimited
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Amlodipine | Udenafil
Number analyzed (Participants) | 26 | 26
cm/sec | -19.9 (145.9) | 63.2 (170.2)

8. Secondary Outcome: Time-averaged Peak Velocity (cm/Sec)
Description: changes in the averaged blood flow (Time-averaged peak velocity) Blood flow in cm/sec 0 - unlimited.
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Amlodipine | Udenafil
Number analyzed (Participants) | 26 | 26
cm/sec | -17.3 (98.6) | 33.4 (123)

9. Secondary Outcome: Dorsal-digital-difference.
Description: The temperature difference between finger tips and dorsum of same hand. range 0 - unlimited in degree celcius.
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: degree celcius.
Arm/Group | Amlodipine | Udenafil
Number analyzed (Participants) | 26 | 26
degree celcius. | -0.7 (3.2) | -1.4 (3.3)

ADVERSE EVENTS:
Time Frame: During 8 weeks while taking a study drug.
Description: As a cross over trial, study participants received both amlodipine and udenafil following each other.
Groups:
- Amlodipine: Adverse effects observed while taking amlodipine in both study arms
- Udenafil: Adverse effects observed while taking udenafil in both study arms
Arm/Group | Amlodipine | Udenafil
Serious Adverse Events (participants affected / at risk) | 0/26 | 2/26
Other Adverse Events (participants affected / at risk) | 14/26 | 19/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amlodipine (N=26) | Udenafil (N=26)
Facial edema (General disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amlodipine (N=26) | Udenafil (N=26)
Facial flushing (General disorders) | 8 (8) | 13 (13)
Facial edema (General disorders) | 4 (4) | 10 (10)
Peripheral edema (General disorders) | 4 (4) | 6 (6)
Headache (General disorders) | 3 (3) | 3 (3)
Blurred vision (Eye disorders) | 2 (2) | 2 (2)
Paresthesia (Nervous system disorders) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Epistaxis (General disorders) | 1 (1) | 0 (0)
Dry mouth (General disorders) | 1 (1) | 0 (0)
Throat irritation (General disorders) | 1 (1) | 0 (0)
Zoster (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No